CLINICAL TRIAL: NCT05972278
Title: A Placebo-Controlled, Phase 1 Study to Investigate the Effect of Obicetrapib on Lipoprotein Metabolism.
Brief Title: Investigating the Effect of Obicetrapib on Lipoprotein Metabolism
Status: Active, not recruiting | Phase: Phase 1 | Type: Interventional
Sponsor: NewAmsterdam Pharma (Industry)
Collaborators: University of Pennsylvania (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: TA-8995-204; The NICE Study (Other: NewAmsterdam Pharma)
Record Dates: First submitted 2023-07-25; First posted 2023-08-02 (Actual); Last update posted 2024-09-19 (Actual); Status verified 2024-09

CONDITIONS: Lipid Metabolism
MeSH Terms: interventions — Tablets

STUDY DESIGN:
Intervention Model Description: This is a phase 1, single-site, double-blind, randomized, placebo-controlled, 2 period, fixed-sequence, pharmacodynamic study in healthy participants meeting the eligibility requirements. Participants will be randomized in a 1:1 ratio to either obicetrapib or matching placebo, and evenly distributed between treatment groups based on their Screening Lp(a) values; ≥ 30 mg/dL vs < 30 mg/dL. LDL-C levels ≥ 100 mg/dL and ≤ 190 mg/dL have been selected for this study as the target population as this is the population of patients targeted for treatment with obicetrapib as an adjunct to statin therapy.
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Masking Description: Double-blind
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Obicetrapib placebo (Placebo Comparator): identical matching placebo
  Interventions: Drug: Obicetrapib
- Obicetrapib 10 mg (Experimental): 10 mg tablets
  Interventions: Drug: Obicetrapib

INTERVENTIONS:
Drug: Obicetrapib — 1 tablet daily
  Other Names: tablets

SUMMARY:
To determine the treatment effect with obicetrapib (10 mg) on the fractional catabolic rate (FCR) of apolipoprotein (apo) B100 in low-density lipoprotein (LDL).

DETAILED DESCRIPTION:
The study population will comprise 20 adults, 18 to 75 years of age, with LDL-C level ≥ 100 and ≤ 190 mg/dL, and in generally good health.

ELIGIBILITY:
Inclusion Criteria:

* Willing to sign the Informed Consent Form.
* Male or female between 18 to 75 years of age.
* Females may be enrolled if they are not pregnant, are not breastfeeding, and do not plan on becoming pregnant during the study.
* Stable weight (± 3 kg) for at least 6 weeks prior to screening.
* Body mass index (BMI) of > 18.5 and ≤ 40 kg/m2 at Screening. BMI is calculated by taking the participants weight in kg and dividing it by the height in meters, squared.
* Participant is judged to be in good health by the Study PI based on medical history, physical examination, vital sign measurements, electrocardiogram (ECG) assessments, and laboratory safety tests performed at Screening and/or prior to administration of the initial dose of study drug.
* Fasting plasma triglyceride level ≤ 400 mg/dL at Screening.
* LDL-C level of ≥ 100 mg/dL and ≤ 190 mg/dL at Screening.

Exclusion Criteria:

* Has taken or plans to take any lipid-lowering medications or medications known to alter lipoprotein metabolism within 4 weeks of Screening, (e.g. statins, fibrates, niacin, cholesterol absorption inhibitors, bile acid-sequestrants, fish oils, PCSK9 inhibitors, red yeast rice, glucocorticoids, and anabolic agents).
* Current, or any previous history of New York Heart Association (NYHA) class III or IV heart failure or left ventricular ejection fraction < 30%.
* Uncontrolled hypertension defined as either systolic blood pressure ≥ 180 mmHg or diastolic blood pressure ≥ 100 mmHg prior to the Baseline visit, taken as the average of triplicate measurements. One triplicate retest will be allowed during the same visit, at which point if the retest result is no longer exclusionary, the participant may be randomized.
* HDL-C > 60 mg/dL if male or >70 mg/dL if female, at Screening.
* An eGFR < 45 mL/min/1.73m2 at the Screening visit or history of end-stage renal disease (ESRD).
* Active liver disease, defined as any known current infectious, neoplastic, or metabolic pathology of the liver; unexplained elevations in alanine aminotransferase (ALT) or aspartate aminotransferase (AST) > 2 x upper limit of normal (ULN); or total bilirubin > 2 x ULN at the and/or Screening visit.
* History of stroke, chronic seizures, or major neurological disorder.
* Participants on thyroid hormone replacement treatment at the time of screening, there is no lower thyroid stimulating hormone (TSH) threshold for entry. The subject must have been on a stable dose of thyroid hormone therapy for ≥ 6 weeks prior to the screening. If TSH levels are undetectable and a change in thyroid hormone therapy is recommended, or if this represents a new diagnosis, then the participant is not eligible. Note: Hypothyroidism is defined as having a TSH > 20% above the local laboratory's upper limit of the normal reference range. One redraw will be allowed if the original TSH value is equal to or less than 40% above the normal reference range at the local laboratory. The participant must meet his criterion upon redraw.
* Participant with a history of neoplastic disease. Note: Participant treated non-melanoma skin carcinoma, and other malignancies which have been successfully treated ≥ 5 years prior to the Screening visit where, in the judgment of both the PI and treating physician, appropriate follow-up has revealed no evidence of recurrence from the time of treatment through the time of the Screening visit.
* Has participated in another investigational drug study within 30 days of Screening

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 22 (Actual)
Dates: Start 2023-12-01 (Actual); Primary Completion 2024-09-26 (Estimated); Study Completion 2024-10-14 (Estimated)

PRIMARY OUTCOMES:
Treatment with obicetrapib (10 mg) on the fractional catabolic rate (FCR) of apolipoprotein (apo) B100 in low-density lipoprotein (LDL). | 8-12 week
  The mean differences (obicetrapib - placebo) in the LDL apoB100 FCR using the baseline measure (no study treatment) compared to the LDL apoB100 FCR of each variable following the Treatment Period.

SECONDARY OUTCOMES:
Treatment with obicetrapib (10 mg) on the production rate (PR) of apolipoprotein(a), or apo(a), in Lp(a). | 8-12 weeks
  The mean differences (obicetrapib - placebo) in the apo(a) in Lp(a) production rate using the baseline measure (no treatment) compared to the apo(a) PR obtained following the Treatment Period.

OTHER OUTCOMES:
Treatment with obicetrapib (10 mg) on the FCR of total apolipoprotein (apo) B100 in plasma. | 8-12 weeks
  The mean difference (obicetrapib - placebo) on the FCR of total apolipoprotein (apo) B100 in plasma using the baseline measure (no treatment) compared to the FCR of apoliprotien (apo) B100 following the Treatment Period.

CONTACTS AND LOCATIONS:
Overall Officials: Archna Bajaj, MD, Principal Investigator — University of Pennsylvania
Locations (1):
- Archna Bajaj, MD, Philadelphia, Pennsylvania, United States

IPD SHARING:
Plan to Share IPD: No